CLINICAL TRIAL: NCT04412096
Title: Aqueous Humor Dynamic Components That Determine Intraocular Pressure Variance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Nebraska (Other); National Eye Institute (NEI) (NIH); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sayoko Moroi, Professor and Chair, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0284; R01EY022124 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma; OHT - Ocular Hypertension
Keywords: aqueous humor dynamics; glaucoma; eye diseases; timolol; latanoprost; Adrenergic beta-Antagonists; Adrenergic Antagonists; Adrenergic Agents; neurotransmitter agents; molecular mechanisms of pharmacological action; physiological effects of drugs; anti-arrhythmia agents; anti-hypertensive agents
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases | interventions — Timolol; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Intervention Model Description: The overall study design is a prospective, open-label, randomized clinical trial with randomized order of 7-day treatments with timolol followed by a washout period and then with latanoprost or vice versa. Participants will undergo two 7-day treatments, with timolol 0.5% (1 drop two times daily) and latanoprost 0.005% (1 drop daily in the evening). The order of timolol and latanoprost will be randomized. The IOP, AHD parameters and IOP fluctuation will be compared in an individual under three conditions: (i) baseline, and after a randomized order of 7-day treatment of (ii) timolol 0.5% 1 drop two times daily and (iii) latanoprost 0.005% 1 drop in the evening separated by a 6-week washout period. The overall time commitment to complete these procedures is three to four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Timolol 0.5% (Experimental): To compare the variation in response to timolol between individuals
  Interventions: Drug: Timolol 0.5% ophthalmic solution
- Latanoprost 0.005% (Experimental): To compare the variation in response to latanoprost between individuals
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: Timolol 0.5% ophthalmic solution — 1 drop BID
  Arms: Timolol 0.5%
Drug: Latanoprost 0.005% Ophthalmic Solution — 1 drop QD
  Arms: Latanoprost 0.005%

SUMMARY:
Glaucoma is a major cause of blindness. The inability to predict a patient's IOP response to medications is a critical barrier for the clinician to consistently provide highly effective IOP-based treatments. Current trial-and-error approaches to glaucoma management are inefficient and have not addressed this barrier as there are no predictive factors for drug response. Our long-term goal is to improve outcomes by identifying biomarkers and environmental factors that profile a patient at risk for glaucoma by age-of-onset, rate of disease progression, "poor response" to treatment, and large IOP fluctuation. Our purpose of this research project is to address this critical barrier by focusing on physiological factors that predict IOP response to drugs.

DETAILED DESCRIPTION:
This proposal responded to PA-18-351 "Human Subjects Mechanistic and Minimal Risk Studies" and qualifies as a clinical trial. The central hypothesis is that variations in IOP response to glaucoma drugs and IOP fluctuation can be predicted by the aqueous humor dynamic (AHD) factors that regulate IOP. This hypothesis will be tested in up to 200 participants with ocular hypertension (OHT) or open-angle glaucoma (OAG). This hypothesis will be tested in two aims: Aim 1, Test the hypothesis that AHD factors predict the IOP drug response; Aim 2, Test the hypothesis that aqueous flow and outflow facility predict IOP fluctuation.

The objective is to determine which AHD factors predict a participant's IOP drug response and IOP fluctuation. The scientific rationale is that AHD parameters (aqueous flow, outflow facility, episcleral venous pressure, and uveoscleral flow) determine drug response and IOP fluctuation.

The primary endpoint is IOP response to glaucoma drugs. Exploratory outcome measures include IOP fluctuation and the AHD measures.

The study population includes participants who have either OHT or OAG. The inclusion and exclusion criteria described in 5.3, Study Population. The goal is to recruit 150-200 participants over 4 years.

All drugs and instruments used in this study have been FDA approved.

Three sites will enroll participants: Mayo Clinic, The Ohio State University, and University of Nebraska Medical Center. All sites have experience and expertise with AHD studies in humans. These study team members have productive collaborations during AHD studies in controls during the prior NIH funding period. There are no sites outside of the United States.

The experimental design is a prospective, open-label, clinical trial with randomized cross over treatment using the topical glaucoma medications, timolol 0.5% and latanoprost 0.005%. Timolol 0.5% is a beta-blocker and will be dosed as one drop two times a day. Latanoprost 0.005% is a prostaglandin analogue and will be dosed as one drop daily in the evening. The treatment order will depend on randomization.

AHD measurements are performed at baseline without glaucoma medications. The AHD measurements include IOP, aqueous humor flow, outflow facility, and episcleral venous pressure. Uveoscleral outflow is calculated. Some participants who are already taking glaucoma medications will be washed out in order to assess baseline AHD measurements. An IOP safety check will be scheduled for those who are washed out of their glaucoma Rx. After baseline AHD measurements, the AHD measurements are repeated after each of the 7-day drug interventions to determine the effect of the drug treatment on AHD variables.

There are six study visits, Visits 1 - 6, that include clinical testing, surveys, and AHD procedures (see 1.2 Schema). Participants will be trained to use the Icare® HOME tonometer to measure IOP outside of clinic to assess IOP fluctuation.

The study design is a prospective, open-label, randomized order of 7-days treatments with timolol 0.5% (1 drop two times daily) followed by a washout period and then with latanoprost 0.005% (1 drop daily in the evening) or vice versa. These are referred to as Tx 1 and Tx 2. IOP safety checks during washout are included for those already taking glaucoma Rx upon entering the study. IOP response will be determined to each of these medications. AHD factors will be determined for both study treatments using tonometry, fluorophotometry, tonography, and episcleral venomanometry. IOP fluctuation will be assessed using the FDA-approved Icare® HOME tonometer. All test procedures and drugs are FDA approved. There are no experimental tests or agents.

Sample sizes and power calculations provide rigor to test the hypothesis.

A REDCap database is populated from data on case report forms (CRF), surveys, and the Icare® HOME tonometer. Data will be analyzed using descriptive statistics of central tendencies and dispersion, and regression methods in order to understand the individual data in the distribution of the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Any self-declared ethnicity-race
* Open-angle with one of the following:

  1. Untreated OHT ≥ 21mmHg
  2. Treated OHT with history of IOP ≥ 21 mmHg on 2 prior clinic visits or IOP ≥ 21 mmHg at screening
  3. Mild-to-moderate stage open-angle glaucoma based on history of untreated IOP ≥ 21 mmHg
* Reliable Humphrey visual field test result within previous 1 year
* Open on gonioscopy within previous 1 year
* At least one eye must be phakic
* Able to cooperate for aqueous humor dynamic procedures
* Able to participate on site over the multi-visit study period
* Contact lenses must be removed before topical fluorescein instillation and remain out until study testing the following day is completed.
* Contact lenses must be removed for the entire duration of the study visits.
* All study medication must be used without contact lenses in the eyes.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* IOP ≥ 38 in study eye(s) or at discretion of the clinician
* Refusal to remove contact lenses
* Advanced visual field loss (MD ≤ -16 dB) or threat to fixation in study eye(s) or at discretion of the clinician
* Study eye(s) with any sign of Fuchs cornea dystrophy as noted clinically with guttae and corneal edema
* Narrow angle of ≤ Shaffer grade 2 for 180 degrees, peripheral synechiae, or peripheral iridotomy in either eye
* History of acute angle closure crisis in either eye
* History of glaucoma incisional surgery (e.g., trabeculectomy, glaucoma drainage implant, Xen gel stent) in study eye(s)
* History of minimally invasive glaucoma surgery (MIGS, e.g., angle surgery, Cypass) in study eye(s)
* History of any cycloablation surgery (e.g., micropulse or diode transcleral or endoscopic cyclophotocoagulation) in study eye(s)
* Study eye cannot have history of any past SLT or ALT glaucoma laser treatments.
* Study eye(s) cannot have any history of refractive surgery
* Study eye(s) cannot have any history of herpetic infection of the cornea
* Study eye(s) cannot have chronic or recurrent inflammatory eye disease
* Study eye(s) cannot have ocular trauma within the past 6 months, other than uncomplicated cornea abrasion
* Study eye(s) cannot have ocular infection in the past 3 months
* Study eye(s) cannot have clinically significant retinal disease that includes proliferative diabetic retinopathy, vein occlusion, cystoid macular edema, wet age-related macular degeneration
* History of intraocular or peri-ocular injections in study eye(s) within 3 months
* History of oral steroid use within 30 days of screening Visit 1
* Any abnormality preventing reliable fluorophotometry (e.g., corneal scarring or severe dry eye with fluorescein staining)
* Serious hypersensitivity to any components of study medications or risk from treatment (e.g., sulfa drug allergy, bradycardia, severe asthma, or emphysema)
* Participants must be on minimum 30-day stable regimen prior to Visit 1 for a systemic medication that may affect IOP (i.e., sympathomimetics, beta-blockers, alpha-adrenergic agonists and blockers, calcium channel blockers, angiotensin converting enzyme inhibitors, etc.). Any change of such medication during the study will result in exclusion.
* Prohibited meds during study: cannabis products, brimonidine 0.025% (Lumify), bimatoprost 0.03% for eyelash growth (Latisse), topical ocular and peri-ocular steroids, oral steroids

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Variation in eye pressures between individuals | measurement after 1 week of treatment
  Eye pressure is a steady state quantitative trait that is measured in mm Hg. Eye pressure is determined by the following physiological factors (units of measure): eye fluid or aqueous humor production (microliters/minute), aqueous humor outflow (microliters/minute), outflow resistance (microliters/minute/mm Hg) and venous pressure (mm Hg) of the eye. All of these physiological factors will be determined under baseline condition and under glaucoma drug treatment.

SECONDARY OUTCOMES:
Variation in aqueous flow between individuals | measurement 1 week after treatment
  Aqueous flow production (microliters/minute) will be determined under baseline condition and under glaucoma drug treatment.
Variation in episcleral venous pressure | measurement 1 week after treatment
  Episcleral venous pressure (mm Hg) of the eye will be determined under baseline condition and under glaucoma drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sayoko Moroi, MD, PhD, Principal Investigator — Professor and Chair
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Man X, Costa R, Ayres BM, Moroi SE. Acetazolamide-Induced Bilateral Ciliochoroidal Effusion Syndrome in Plateau Iris Configuration. Am J Ophthalmol Case Rep. 2016 Oct;3:14-17. doi: 10.1016/j.ajoc.2016.05.003. Epub 2016 May 17. PMID 29226268
- [Derived] Kazemi A, Reitinger JC, Toris CB, Gulati V, Fan S, Reed DM, Moroi SE, Sit AJ. Aqueous Humor Dynamics Changes and Predictors of IOP Response to Latanoprost in Healthy Subjects. J Glaucoma. 2025 Dec 1;34(12):1056-1064. doi: 10.1097/IJG.0000000000002585. Epub 2025 May 9. PMID 40341017

DOCUMENTS (1):
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04412096/ICF_001.pdf